CLINICAL TRIAL: NCT03278639
Title: Randomized, Blind, Controlled Clinical Trial to Assess the Efficacy and Safety or Rhythmic Auditory Stimulation (RAS) for Gait and Balance Disorders in Parkinson's Disease
Brief Title: Efficacy and Safety or Rhythmic Auditory Stimulation (RAS) for Gait and Balance Disorders in Parkinson's Disease
Acronym: ERA-EP2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We could not fund the study
Sponsor: Pontifical Catholic University of Argentina (Other)
Collaborators: National Council of Scientific and Technical Research, Argentina (Other Government); Hospital Nacional Profesor Alejandro Posadas (Other); University of Buenos Aires (Other)
Responsible Party: Principal Investigator, Santiago Perez Lloret, MD PhD CPI, Pontifical Catholic University of Argentina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERAEP2
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease
Keywords: gait disorders; balance disorders; music; tango; rhythmic auditory stimulation; health-related quality of life
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation | interventions — Kinesiology, Applied

STUDY DESIGN:
Intervention Model Description: randomized, prospective, blind, controlled clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both investigators taking care of patients and outcomes assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythmic auditory stimulation (Experimental): Each patient will receive training for 4 weeks, 3 times per week. Each training session will last 30 minutes. Training will be performed by music therapists board-certified in RAS.
  Interventions: Behavioral: Rhythmic Auditory Stimulation
- Kinesiology (Active Comparator): Each patient will receive training for 4 weeks, 3 times per week. Each training session will last 30 minutes. Training will be performed by board-certified kinesio therapists. The objectives of the training sessions will match those of RAS.
  Interventions: Behavioral: Kinesiology

INTERVENTIONS:
Behavioral: Rhythmic Auditory Stimulation — Training will be directed to ameliorate gait and balance
  Arms: Rhythmic auditory stimulation
Behavioral: Kinesiology — Training will be directed to ameliorate gait and balance
  Arms: Kinesiology

SUMMARY:
Gait deficits are among the most characteristic and most functionally debilitating signs of the motor neuropathology of Parkinson's disease (PD). Rhythmic Auditory Stimulation (RAS) is a technique by which a series of auditory stimuli are presented at a fixed rhythm, so that patients have to synchronize their movements to the rhythms. In this study, auditory stimuli will be constituted by Tango musical pieces, which tempo is modified to adapt to patients' walking cadence. Previous results suggested that RAS can increase Tinetti's gait and balance and may also improve Health-Related Quality of Life. This will be a randomized, blind, controlled clinical trial to further assess RAS efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definitive or probable PD diagnosis
* Gait disorders (MDS-UPDRS #2.12 =1)
* Patients that can be reasonably expected to remain in ON-state during training sessions.

Exclusion Criteria:

* Previous use of RAS or kinesiology
* MMSE >= 24
* BDI >= 17
* Patients having undergone PD surgical treatments.
* Patients with auditory or visual handicaps

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
change from baseline in Tinetti scale total score | 4 weeks

SECONDARY OUTCOMES:
change from baseline in Tinetti scale Gait score | 4 weeks
change from baseline in Tinetti scale Balance score | 4 weeks
change from baseline in Tinetti scale total score | 6 months
  training will last for the first 4 weeks. Assessments will be also performed at Month 6 to check lasting effects.
change from baseline in Timed Up & Go test (TUG) | 4 weeks
change from baseline in PDQ-39 scores | 4 weeks
  PDQ-39 is a PD-specific scale for Health-related Quality of Life
change from baseline in MDS-UPDRS score | 4 weeks
  MDS-UPDRS is a measure of disease severity
change from baseline in Beck Depression Index (BDI) | 4 weeks
change from baseline in MMSE (Mini-Mental State Examination) | 4 weeks
  MMSE is a measure of cognitive impairment
change from baseline in Fall diary | 4 weeks
  patients will have to indicate the number of daily falls over a 15-d period

OTHER OUTCOMES:
change from baseline in PD CRS | 4 weeks and 6 months
  Parkinson's Disease Cognitive Rating Scale (PD CRS) measures cognitive performance
change from baseline in DRS | 4 weeks and 6 months
  Dementia Rating Scale (DRS) measures cognitive performance
change from baseline in TUG | 6 months
change from baseline in PDQ-39 | 6 months
change from baseline in MDS-UPDRS | 6 months
change from baseline in BDI | 6 months
change from baseline in MMSE | 6 months
change from baseline in fall diary | 6 months

IPD SHARING:
Plan to Share IPD: No